CLINICAL TRIAL: NCT04289922
Title: Cross-cultural Adaption and Validation of the Norwegian VISA-G Questionnaire for Patients With Hip Pain
Brief Title: Validation of the Norwegian VISA-G Questionnaire
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Håkon Sveinall, Principal Investigator, Oslo University Hospital
Other Study IDs: REK 2019/428 A
Record Dates: First submitted 2020-02-21; First posted 2020-02-28 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Hip Pain Chronic; Hip Bursitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to translate, cross-cultural adapt and validate the Norwegian VISA-G (VISA-N-G) questionnaire. The study will test the psychometric properties for the VISA-N-G in terms of test-retest reliability, internal consistency, construct validity and responsiveness.

DETAILED DESCRIPTION:
The Victorian Institute of Sport Assessment-Gluteal Questionnaire (VISA-G) questionnaire have already been developed and used as a measurement tool in research on English speaking Greater trochanteric pain syndrome (GTPS) populations.

The aim of this study is to translate, cross-cultural adapt and validate the Norwegian VISA-G (VISA-N-G) questionnaire.

The translation of the original VISA-G into Norwegian has been done following the official guidelines.

The patients will be recruited from the outpatient clinic at the Department of Physical Medicine and Rehabilitation, Oslo University Hospital and will follow the ordinary patient care.

After given written consent, patients will be asked to fill out the following Norwegian questionnaires: VISA-N-G, Harris Hip Score (HHS), Oswestry disability index (ODI) and a numeric rating scale (NRS) for assessment of pain intensity. The aforementioned questionnaires will be used to test the construct validity with various hypothesis at baseline. Within one week the investigators will ask the patients to fill out the VISA-N-G once more to test the test-retest reliability.

To investigate responsiveness the patient will be asked to fill out the VISA-N-G together With HHS, ODI, NRS and a 11-Point Global Rating of Change scale (GROC) after seven weeks. Responsiveness will be tested with various hypothesis and measured by the area under the receiver operating characteristics curve (ROC).

ELIGIBILITY:
Inclusion Criteria:

* Hip pain
* Ability to read and write Norwegian
* > 18 years old

Exclusion criteria:

* Not able to read and write Norwegian
* < 18 years old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients included in our project is referred to the Department of Physical Medicine and Rehabilitation through a primary contact in the primary health care i.e. medical doctors, manual therapists or chiropractors, or from other doctors within the specialist healthcare settings for example a rheumatologists or orthopaedic surgeons. The investigators will record information on age, gender, education and work status in addition to data from the included questionnaires.
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
VISA-N-G | Baseline, 1 week, 7 weeks.
  The Victorian Institute of Sport Assessment-Gluteal Questionnaire (VISA-G) questionnaire have already been developed and used as a measurement tool in research on English speaking GTPS populations.The VISA-G questionnaire is based on other Health-related patient-reported outcomes (HR-PROs) from Victorian Institute of Sports tendon study Group. The investigators will test the construct validity with two other HR-PROs (Harris Hip Score and Oswestry disability index). To investigate test-retest reliability, the patients will fill out a second VISA-N-G one week after baseline. To test responsiveness, the patients will fill out VISA-N-G 7 weeks after baseline together with the two other HR-PROs, and a Global Rating of Change scale.

SECONDARY OUTCOMES:
Harris Hip Score | Baseline, 7 weeks
  Harris Hip Score (HHS) is an HR-PROs questionnaire used for assessing outcome after total hip replacement, femoral neck fractures and osteoarthritis. It is expected to take 5 minutes to complete and is based on 10 items. It is scored from 0 to 100, where 100 is the best outcome, <70 is considered a poor result. HHS has shown to be a responsive measure and shows a strong correlation in the physical domain of The short form Health survey (SF36) and high correlation to the Nottingham Health Profile.
Oswestry disability index | Baseline, 7 weeks
  Oswestry disability index (ODI) is a widely used HR-PROs used for spinal disorders. Its asking about the patients perceived disability and is scored from 0 to 100%, where 0% indicates no disability and 100% indicates most disability. ODI is cross-cultural adapted into Norwegian and psychometric properties was concluded acceptable for assessing self-reported functional status of Norwegian-speaking patients with low back pain.
Numeric rating scale | Baseline, 7 weeks
  In a Numeric rating scale (NRS) the patients rate their pain intensity between 0 and 10. Zero represents "no pain at all" and 10 represents "the worst pain ever possible". NRS correlates highly to other pain assessment tools. A change of two points is detected as being clinically significant. In this project the investigator will ask for the patient's current pain, average pain the last week, worst pain last week, and least pain last week.
Global Rating of Change scale | Baseline, 7 weeks
  A Global Rating of Change scale (GROC) scale is designed to quantify a patient's improvement or worsening over time, the scale ask about the current and previous health status and then calculates the difference. The scale is "global" and allows the patient themselves to subjectively decide their health status. Scales between 7 and 11 seems to be the compromise between patient preference, adequate discriminative ability and test-retest reliability. The investigator will use an 11-point scale from - 5 to 5 where - 5 = worsening, 0 = unchanged and 5 = completely recovered. An 11-point scale has shown test-retest reliability with ICC 0.90, minimum detectable change of 0.45 points and minimally clinically important change 2 points.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne B Johnsen, PT, MSc, PhD, Study Director — Oslo University Hospital, Department of Physical Medicine and Rehabilitation
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Background] Fearon AM, Ganderton C, Scarvell JM, Smith PN, Neeman T, Nash C, Cook JL. Development and validation of a VISA tendinopathy questionnaire for greater trochanteric pain syndrome, the VISA-G. Man Ther. 2015 Dec;20(6):805-13. doi: 10.1016/j.math.2015.03.009. Epub 2015 Apr 2. PMID 25870117
- [Background] Mokkink LB, Terwee CB, Patrick DL, Alonso J, Stratford PW, Knol DL, Bouter LM, de Vet HC. The COSMIN checklist for assessing the methodological quality of studies on measurement properties of health status measurement instruments: an international Delphi study. Qual Life Res. 2010 May;19(4):539-49. doi: 10.1007/s11136-010-9606-8. Epub 2010 Feb 19. PMID 20169472
- [Background] Nilsdotter A, Bremander A. Measures of hip function and symptoms: Harris Hip Score (HHS), Hip Disability and Osteoarthritis Outcome Score (HOOS), Oxford Hip Score (OHS), Lequesne Index of Severity for Osteoarthritis of the Hip (LISOH), and American Academy of Orthopedic Surgeons (AAOS) Hip and Knee Questionnaire. Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S200-7. doi: 10.1002/acr.20549. No abstract available. PMID 22588745
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Derived] Sveinall H, Wenstad PK, Fearon AM, Skyttemyr G, Thornes E, Skaara HE, Juel NG, Brox JI, Roe C, Johnsen MB. The reliability and validity of the Norwegian version of the Victorian Institute of Sports Assessment for gluteal tendinopathy questionnaire (VISA-G-Norwegian) for patients with greater trochanteric pain syndrome. BMC Musculoskelet Disord. 2023 Sep 29;24(1):769. doi: 10.1186/s12891-023-06901-0. PMID 37770944